CLINICAL TRIAL: NCT00005096
Title: Docetaxel Followed by Radical Prostatectomy in Patients With High Risk Localized Prostate Cancer
Brief Title: Docetaxel in Treating Patients With Stage II or Stage III Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rhone-Poulenc Rorer (Industry)
Responsible Party: Principal Investigator, Mary-Ellen Taplin, MD, Taplin, Mary-Ellen, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99-193; P30CA006516 (NIH); DFCI-99193; NCI-G00-1757
Record Dates: First submitted 2000-04-06; First posted 2004-03-04 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage II prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel (Experimental): Docetaxel given via iv at determined dose once a week for 4 weeks
  Interventions: Drug: docetaxel

INTERVENTIONS:
Drug: docetaxel
  Other Names: Taxotere

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of docetaxel in treating patients who have stage II or stage III prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the pathologic complete response rate to docetaxel in patients with high risk stage II or III prostate cancer. II. Determine the toxicity of this treatment in these patients. III. Correlate clinical measures of response (e.g., symptoms, physical exam, serum PSA, and endorectal MRI) with pathologic response to this treatment in these patients.

OUTLINE: Patients receive docetaxel IV over 30 minutes weekly for 4 weeks. Treatment continues for 2-6 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 19-45 patients will be accrued for this study over 18 months.

ELIGIBILITY:
Eligibility Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Potential candidate for radical prostatectomy
* Any of the following:

  * Clinical stage T3 patients
  * Serum PSA at least 20 ng/mL
  * Gleason score 8-10
  * Clinical T2 disease and either of the following:

    * MRI evidence of seminal vesicle involvement
    * Gleason 4+3 cancer with either 5 or 6 biopsies positive
* CALGB 0-1
* WBC greater than 3,000/mm3
* Hematocrit greater than 30%
* Platelet count greater than 100,000/mm3
* SGOT, total bilirubin within normal limits
* Signed Informed consent

Exclusion Criteria:

* No prior hormones, radiation or chemotherapy for prostate cancer
* Evidence of serious active infection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 1999-12 (Actual); Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Complete Response Rate | 2 Months, 6 Months
  Wilcoxon Signed Rank Test

SECONDARY OUTCOMES:
Percentage of Participants with mild to moderate toxicity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Ellen Taplin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No